CLINICAL TRIAL: NCT05287412
Title: Long-Term Outcomes After the Multisystem Inflammatory Syndrome in Children
Acronym: MUSIC
Status: Active, not recruiting | Type: Observational
Sponsor: Carelon Research (Other)
Responsible Party: Sponsor
Other Study IDs: G20479
Record Dates: First submitted 2022-02-09; First posted 2022-03-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Multisystem Inflammatory Syndrome in Children (MIS-C)
Keywords: COVID
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood or saliva that is collected for future whole genome sequencing will be requested as optional at any time that the patient is undergoing a clinical laboratory draw in participants who provide consent for this testing. To better understand the genetic variation within the heterogenous MIS-C population, blood or saliva samples from the biological parents of MIS-C patients will also be requested as optional. Samples from parents will also be stored at the similar venue for future whole genome sequencing. In addition, the study investigators expect to collaborate with centers or networks that are collecting research samples on these patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Multi-system Inflammatory Syndrome in Children (MIS-C) is a new condition related to COVID-19, the study investigators are still learning about its causes, effects, and long-term impact. "Long-Term Outcomes after the Multisystem Inflammatory Syndrome In Children", the Coronavirus MUSIC Study, is a research study funded by NIH and the National Heart, Lung, and Blood Institute. The study investigators hope to enroll at least 900 young people with MIS-C at children's medical centers in the U.S. and Canada. This research study will help us learn more about MIS-C and its effects on the long-term health of children.

DETAILED DESCRIPTION:
This study is an observational cohort study that will use routinely collected clinical and cardiac (EKG, echocardiogram, Cardiac MRI, exercise testing) data to assess the association between MIS-C and cardiac outcomes within the first year after hospital discharge. Research funding will be available for EKGs, echocardiograms and MRIs in protocol windows that are not ordered by primary caregivers. The principal goal is to determine the spectrum and early time course of coronary artery involvement, LV systolic function, and arrhythmias or conduction system abnormalities, and, using these data, to define associated clinical and laboratory factors. The study investigators planned to include all eligible patients, including retrospective cases beginning January 1, 2020, with follow-up (in-person or telehealth) to up within one year and annual medical history forms until up to 5 years have elapsed since illness onset. Because many patients will have been identified by retrospective review, the study team will obtain consent at different times in their illness course. For this reason, it may be hard to reach some patients and their families. Waiver of consent will be obtained after three attempts have been made to locate the patient and family without success, as well as for the rare child who dies before informed consent can be obtained. The study investigators will include a HIPAA-compliant cryptographic algorithm to create a sharable "hashed" identifier from patient information. If blood work for research purposes is added on to usual clinically indicated blood work during follow-up visits, this will be covered by other informed consent forms.

ELIGIBILITY:
Inclusion Criteria:

1. Age <21 years.
2. Fever ≥38°C for ≥24 hours, or report of subjective fever lasting ≥24 hours.
3. Laboratory evidence of inflammation, including, but not limited to, one or more of the following: an elevated CRP, ESR, fibrinogen, procalcitonin, d-dimer, ferritin, LDH, or IL-6, elevated neutrophils, reduced lymphocytes and low albumin.
4. Evidence of clinically severe illness requiring hospitalization, with multisystem (≥2) organ involvement, based on clinical judgment from record review, discharge diagnosis, laboratory or diagnostic tests. Organ system involvement includes but is not limited to cardiac, renal, respiratory, hematologic including coagulopathy, gastrointestinal including liver, dermatologic or neurological.
5. Positive for current or recent SARS-CoV-2 infection by RT-PCR, serology, or antigen test; or COVID-19 exposure within the 4 weeks prior to the onset of symptoms

Exclusion Criteria:

* No plausible alternative diagnosis, such as bacterial sepsis, murine typhus, staphylococcal or streptococcal shock syndromes

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children and young adults <21 years with Multisystem Inflammatory Syndrome in Children associated with COVID-19 (MIS-C) at a participating hospital
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
worst-ever LV ejection fraction | hospital admission through 5 years post-hospitalization
  worst left ventricular (LV) ejection fraction from core lab echo read during MUSIC study
worst-ever maximum z score of the proximal LAD or RCA | hospital admission through 5 years post-hospitalization
  worst maximum z-score of the proximal left anterior descending coronary artery (LAD) or right coronary artery (RCA) from core lab echo read; z-scores to be calculated via Boston z-score calculator (primary) and Pediatric Heart Network z-score calculator (secondary); higher z-scores are worse

SECONDARY OUTCOMES:
Occurrence of a proximal LAD or RCA z score of ≥2.5 on any echocardiogram | hospital admission through 5 years post-hospitalization
  proximal left anterior descending coronary artery (LAD) or right coronary artery (RCA) ≥2.5 from any core lab echo read
Occurrence of aneurysms by Japanese Ministry of Health criteria | hospital admission through 5 years post-hospitalization
  Occurrence of aneurysms by Japanese Ministry of Health criteria applied to core lab echo reads
Individual z scores for LMCA, RCA and LAD | hospital admission through 5 years post-hospitalization
  Individual z scores for left main coronary artery (LMCA), right coronary artery (RCA) and proximal left anterior descending coronary artery (LAD) as per core lab echo reads; higher z-scores are worse
LVEDV z score | hospital admission through 5 years post-hospitalization
  left ventricular (LV) size as measured by left ventricular end-diastolic volume (LVEDV) z score
LVEF | hospital admission through 5 years post-hospitalization
  left ventricular (LV) function as measured by left ventricular ejection fraction (LVEF)
LVSF | hospital admission through 5 years post-hospitalization
  left ventricular (LV) function as measured by left ventricular shortening fraction (LVSF)
The percentage of patients who had LV ejection of <55%, and further categorization of 45-54% (i.e., mildly depressed systolic function), 35-44% (moderately depressed systolic function) and <35% (severely depressed systolic function) on any echocardiogram | hospital admission through 5 years post-hospitalization
  The percentage of patients who had left ventricular (LV) ejection of <55%, and further categorization of 45-54% (i.e., mildly depressed systolic function), 35-44% (moderately depressed systolic function) and <35% (severely depressed systolic function) on any echocardiogram read by the core lab
LV strain (global longitudinal strain from apical view and global circumferential strain from parasternal short-axis view) | hospital admission through 5 years post-hospitalization
  left ventricular (LV) strain (global longitudinal strain from apical view and global circumferential strain from parasternal short-axis view) on core lab echo read
Qualitative assessment of RV systolic function | hospital admission through 5 years post-hospitalization
  Qualitative assessment of right ventricular (RV) systolic function on core lab echo read
Qualitative assessment of RV global longitudinal strain | hospital admission through 5 years post-hospitalization
  Qualitative assessment, if possible, of right ventricular (RV) global longitudinal strain on core lab echo read
Presence and degree of mitral and aortic regurgitation | hospital admission through 5 years post-hospitalization
  Presence and degree of mitral and aortic regurgitation on echo core lab read
LV diastolic function, i.e., tissue Doppler imaging and mitral valve (MV) inflow | hospital admission through 5 years post-hospitalization
  left ventricular (LV) diastolic function, i.e., tissue Doppler imaging and mitral valve (MV) inflow on echo core lab read
Presence and size of pericardial effusion | hospital admission through 5 years post-hospitalization
  Presence and size of pericardial effusion on echo core lab read
The occurrence of arrhythmias and conduction system disturbances by in-hospital monitoring, electrocardiograms, and exercise testing at 3 months in those with a history of ≥moderate systolic dysfunction when age and maturity permit | 3 months post-discharge
  The occurrence of arrhythmias and conduction system disturbances by in-hospital monitoring, electrocardiograms, and exercise testing at 3 months in those with a history of ≥moderate systolic dysfunction when age and maturity permit
MRI LVEF | hospital admission through 5 years post-hospitalization
  LVEF on MRI core lab read
MRI RVEF | hospital admission through 5 years post-hospitalization
  RVEF on MRI core lab read
valvar regurgitation | hospital admission through 5 years post-hospitalization
  valvar regurgitation on MRI core lab read
myocardial late gadolinium enhancement (LGE) | hospital admission through 5 years post-hospitalization
  percent with and distribution of myocardial late gadolinium enhancement (LGE) on MRI core lab read
abnormal T2-weighted imaging | hospital admission through 5 years post-hospitalization
  percent abnormal T2-weighted imaging on MRI core lab read
elevated T2 | hospital admission through 5 years post-hospitalization
  percent with elevated T2 on MRI core lab read
elevated native T1 | hospital admission through 5 years post-hospitalization
  percent with elevated native T1 on MRI core lab read
elevated extracellular volume fraction | hospital admission through 5 years post-hospitalization
  percent with elevated extracellular volume fraction on MRI core lab read
coronary artery dilation | hospital admission through 5 years post-hospitalization
  percent with coronary artery dilation on MRI core lab read
CMR abnormal, equivocal, or negative | hospital admission through 5 years post-hospitalization
  final interpretation of CMR as abnormal, equivocal, or negative (i.e., no abnormal or equivocal findings) on MRI core lab read
Other organ abnormalities by medical history: Immunologic, rheumatologic, renal, pulmonary, hematologic, gastrointestinal, dermatologic or neurologic | hospital admission through 5 years post-hospitalization
  percent with other organ abnormalities by medical history: Immunologic, rheumatologic, renal, pulmonary, hematologic, gastrointestinal, dermatologic or neurologic
CRP | hospital admission through 5 years post-hospitalization
  C-Reactive Protein (CRP) as a laboratory marker of inflammation
Admission to ICU | hospital admission through 5 years post-hospitalization
  percent with admission to ICU
Maximal vasoactive inotrope score | from MIS-C hospital admission to MIS-C hospital discharge
  Maximal vasoactive inotrope score
Hospital length of stay | from MIS-C hospital admission to MIS-C hospital discharge
  Hospital length of stay
Symptom duration | hospital admission through 5 years post-hospitalization
  Symptom duration
Major medical events | hospital admission through 5 years post-hospitalization
  percent with major medical events (e.g., stroke, need for extracorporeal therapies such as renal replacement therapy, plasma exchange, ECMO, VAD)
Mortality | hospital admission through 5 years post-hospitalization
  Percent mortality
Global Health - FSS | hospital admission through 5 years post-hospitalization
  Global Health as measured by Functional Status Score [FSS]: range 6-30, lower is better
Global Health - PROMIS | hospital admission through 5 years post-hospitalization
  Global Health as measured by Parent-Reported Outcomes Measurement Information Systems [PROMIS] Instrument: range 7-35, higher is better

CONTACTS AND LOCATIONS:
Locations (33):
- United States (32):
  - University of Alabama, Tuscaloosa, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Valley Children's Healthcare and Hospital, Madera, California
  - UC San Diego, Rady Children's Hospital, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - The Nemours Foundation, Wilmington, Delaware
  - Children's National Hospital, Washington D.C., District of Columbia
  - Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Chldren's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert Lurid Children's Hospital of Chicago, Chicago, Illinois
  - Riley Children's Hospital, Indianapolis, Indiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - CS Mott Children's Hospital/University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Morgan Stanley Children's Hospital of New York, New York, New York
  - Cohen Children's Medical Center, Queens, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke Children's Hospital and Health Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Dell Medical Center, Austin, Texas
  - Children's Medical Center of Dallas - UT Southwestern Medical Center, Dallas, Texas
  - Baylor /Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Medical College of Wisconsin/Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lang SM, Truong DT, Powell AJ, Kazlova V, Newburger JW, Awerbach JD, Binka E, Bradford TT, Cartoski M, Cheng A, DiLorenzo MP, Dionne A, Dorfman AL, Elias MD, Garuba O, Gerardin JF, Hasbani K, Jone PN, Lam CZ, Misra N, Morgan LM, Nutting A, Patel JK, Robinson JD, Schuchardt EL, Sexson Tejtel K, Singh GK, Slesnick TC, Trachtenberg F, Taylor MD; MUSIC Study Investigators. CMR Findings in the Long-Term Outcomes After Multisystem Inflammatory Syndrome in Children (MUSIC) Study. Circ Cardiovasc Imaging. 2025 Sep;18(9):e017420. doi: 10.1161/CIRCIMAGING.124.017420. Epub 2025 Apr 4. PMID 40181776